CLINICAL TRIAL: NCT00457600
Title: ParentLink: Better and Safer Emergency Care for Children
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: South Shore Hospital (Other)
Other Study IDs: CHB-R01HS014947
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-01

CONDITIONS: Otitis Media; Urinary Tract Infection; Asthma; Head Injury
Keywords: information technology; emergency department; medication error; quality of care; patient-centered care
MeSH Terms: conditions — Otitis Media; Urinary Tract Infections; Asthma; Craniocerebral Trauma; Emergencies

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: patient-driven health IT product

SUMMARY:
The emergency department (ED) constitutes a high-risk environment for errors and poor quality of care. Pediatric patients are at increased risk of medical errors. We postulate that implementation of a patient-centered health information technology - ParentLink - can address system-level deficiencies and the unique "just-in-time" information needs of ED physicians and the parents of ill children. The proposed work delivers an innovative product - an electronic interface linked to a pediatric knowledge base that integrates parent-derived data with best practices for safe and effective emergency care across common pediatric disease conditions: otitis media, urinary tract infections, asthma, and head trauma. The study has two aims, the first of which addresses critical gaps in data capture: to evaluate the completeness and accuracy of information on symptoms, disease condition, medications and allergies generated by parents using ParentLink versus information documented by ED physicians and nurses, using structured telephone interviews as a gold standard. The second aim measures the ParentLink's impact on ED patient safety and quality, specifically: a) the error rate for ordering and prescribing of medications during ED care, and b) the percent of ED visits that adhere to national evidence-based guidelines. Parentlink will be rigorously evaluated in a clinical trial at two diverse ED sites and will use a sequential, non-randomized observational design with two intervention and two control periods to measure the effects of ParentLink on data capture and safety and quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 12 years with head trauma
* Age less than 12 years with ear pain
* Ages less than 12 years with concern for UTI
* 1 year - 12 years with asthma history and respiratory chief complaint
* 3 months - 2 years with fever
* Parent speaks English or Spanish
* Triage status is non-emergent

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000
Dates: Start 2005-06; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C Porter, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts